CLINICAL TRIAL: NCT03570541
Title: Improving Perioperative Pain Management for Laparoscopic Surgery Due to Colon Cancer Using the Ultrasound-guided Transmuscular Quadratus Lumborum Block. A Double Blind, Randomized, Placebo Controlled Trial.
Brief Title: TQL-block for Laparoscopic Hemicolectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJ-663; 2017-005200-96 (EudraCT Number)
Record Dates: First submitted 2018-05-15; First posted 2018-06-27 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain
Keywords: Colon cancer; nerve block; ultra-sound; opioids; surgical stress
MeSH Terms: conditions — Pain, Postoperative; Colonic Neoplasms | interventions — Ropivacaine; Acetaminophen; Analgesia, Patient-Controlled; Morphine; Sodium Chloride; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Active bilateral ultrasound-guided transmuscular quadratus lumborum (TQL) block. 60 mL ropivacaine 0,375% single shot.
  Every six hours postoperative, all patients are administered 1 g of acetaminophen.
  In both arms morphine will be administered IV as part of a patient controlled analgesia (PCA)-pump regimen or additionally after contact with the nursing staff as it is the standard treatment.
  On the day of surgery, postop day 1+2 and day 10-14, all patients will have blood samples taken for immunological analysis.
  On the day of surgery, postop day 1+2 and day 10-14, all patients are asked to fill out a Quality of recovery-15 questionaire.
  Before surgery, and 3, 6 and 24 hours postop. All patients are tested for orthostatic hypotension.
  Interventions: Drug: Ropivacaine; Drug: Acetaminophen; Device: Patient controlled analgesia; Drug: Morphine; Diagnostic Test: Blood samples; Behavioral: Quality of recovery-15 questionaire; Diagnostic Test: Orthostatic hypotension
- Placebo (Placebo Comparator): Placebo bilateral ultrasound-guided transmuscular quadratus lumborum (TQL) block. 60 mL saline single shot.
  Every six hours postoperative, all patients are administered 1 g of acetaminophen.
  In both arms morphine will be administered IV as part of a patient controlled analgesia (PCA)-pump regimen or additionally after contact with the nursing staff as it is the standard treatment.
  On the day of surgery, postop day 1+2 and day 10-14, all patients will have blood samples taken for immunological analysis.
  On the day of surgery, postop day 1+2 and day 10-14, all patients are asked to fill out a Quality of recovery-15 questionaire.
  Before surgery, and 3, 6 and 24 hours postop. All patients are tested for orthostatic hypotension.
  Interventions: Drug: Acetaminophen; Device: Patient controlled analgesia; Drug: Morphine; Drug: Saline; Diagnostic Test: Blood samples; Behavioral: Quality of recovery-15 questionaire; Diagnostic Test: Orthostatic hypotension

INTERVENTIONS:
Drug: Ropivacaine — 30 mL ropivacaine 0,375% administered on each side as bilateral TQL blocks
  Arms: Active
Drug: Acetaminophen — Every six hours postoperative, all patients are administered 1 g of acetaminophen.
Device: Patient controlled analgesia — PCA-pump with IV-Morphine. 5 mg administered per bolus. Lock-out time and max. dosage standardized.
Drug: Morphine — intravenously administered morphine via PCA-pump
Drug: Saline — 30 ml saline 0,375% administered on each side as bilateral TQL blocks
  Arms: Placebo
Diagnostic Test: Blood samples — On the day of surgery, postop day 1+2 and day 10-14, all patients will have blood samples taken for immunological analysis
Behavioral: Quality of recovery-15 questionaire — On the day of surgery, postop day 1+2 and day 10-14, all patients are asked to fill out a short questionaire.
Diagnostic Test: Orthostatic hypotension — Before surgery, and 3, 6 and 24 hours postop. All patients are tested for orthostatic hypotension.

SUMMARY:
Every year 350 patients undergo surgery due to colorectal cancer at Zealand University Hospital, Roskilde. The majority of the surgeries are performed using a minimal invasive laparoscopic technique where the bowl anastomosis is either hand sown or stapled. The procedure is performed, while the patient is under general anaesthesia.

An observational prospective survey from 2016-17 of sixty patients undergoing hemicolectomy at Zealand University Hospital, Roskilde has shown, that even though the patients are subjected to a multimodal analgesic regimen, a substantial amount of opioids are being administered during the first 24 hours post surgery; i.e. 51.91 mg ± 36.22 mg (Mean ± SD) of oral morphine equivalents. Sixty-five percent of the patients receive opioids at the PACU. Their maximum pain score at the PACU is registered, using a numerical rating scale of 0-10, as 3.28 ± 2.65 (Mean ± SD). So it is obvious that there is room for improvement and a reduction in the use of postoperative opioids. Thus, there is a clearly defined research problem to explore.

Currently ultrasound-guided nerveblocks are not part of the multimodal analgesic regimen.

The primary aim of this study is to investigate the efficacy of the ultrasound-guided bilateral transmuscular quadratus lumborum block on reducing postoperative opioid consumption.

DETAILED DESCRIPTION:
Every year 350 patients undergo surgery due to colorectal cancer at Zealand University Hospital, Roskilde. The vast majority of the patients has to have part of their colon removed, a so-called hemicolectomy. The majority of the surgeries are performed using a minimal invasive laparoscopic technique where the bowl anastomosis is either hand sown or stapled. The procedure is performed, while the patient is under general anaesthesia using a continuous intravenous (iv.) infusion of propofol and remifentanil to keep the patient asleep. As postoperative pain management the patients receive IV. paracetamol, IV. sufentanil (30 minutes prior to surgery) and local would infiltration.

At the post anaesthesia care unit (PACU) the patients are offered paracetamol and morphine as pain management. An observational prospective survey from 2016-17 of sixty patients undergoing hemicolectomy at Zealand University Hospital, Roskilde has shown, that even though the patients are subjected to a multimodal analgesic regimen as described, a substantial amount of opioids are being administered during the first 24 hours post surgery; i.e. 51.91 mg ± 36.22 mg (Mean ± SD) of oral morphine equivalents. Sixty-five percent of the patients receive opioids at the PACU. Their maximum pain score at the PACU is registered, using a numerical rating scale of 0-10, as 3.28 ± 2.65 (Mean ± SD). So it is obvious that there is room for improvement and a reduction in the use of postoperative opioids. Thus, there is a clearly defined research problem to explore.

Surgical technique:

The procedure is performed as a standard 4 port laparoscopic or robot-assisted technique with a vessel first dissection approach. The principles of complete mesocolic excision with is the standard procedure. The extraction site is for the right side and transverse colon through an upper transverse incision and for the left side and rectum through a pfannenstiel incision.

Anaesthesia and postoperative pain management:

The laparoscopic hemicolectomy is performed with the patient under general anaesthesia. As the surgery ends the surgeon injects local would infiltration in the laparoscopic port entries. Around 30 minutes prior to emergence the anaesthetic nurse injects iv. sufentanil (synthetic morphine), often around 0.3 μg/kg and 1g of iv. paracetamol. At the PACU a nurse will administer iv. morphine or sufentanil or oral morphine, when needed. The postoperative pain management continues at the surgical ward, where morphine is administered when needed. Paracetamol 1 gram x 4 daily is administered until discharge.

Side effects of current treatment:

The use of morphine can cause severe side effects, including nausea and vomiting, bowl paralysis, urine retention, sleep disturbances and respiratory depression. These side effects can delay mobilisation after surgery, increase the risk of complications and worst of all be fatal.

Recent research indicates a connection between immunologic and stress related reactions in relation to surgery and the development of cancer metastasis. It has already been shown, that a minimal invasive surgical technique, laparoscopic vs. open surgery, improves the postoperative immunologic response. A recent meta-analysis shows that perioperative regional anaesthesia/analgesia improves survival in cancer patients, which can be related to a reduction in metastasis due to a reduced surgical stress response. This indicates, that there are multiple advantages in offering an opioid sparing pain management, that also reduces the stress response related to surgery. The short term advantage being a reduction in postoperative opioid consumption, opioid-related side effects and postoperative pain score and possibly a long-term advantage of fewer cancer recurrences.

Ultrasound-guided nerve blocks:

With regards to the side effects related to the current treatment it has been of the upmost interest to develop new techniques to manage postoperative pain and a at the same time reduce surgical stress. Associate Professor and head of research at The Department of Anaesthesiology and Intensive Care, Jens Børglum, has in collaboration with other international peripheral nerve block experts developed several different abdominal nerve blocks that are described in both cadaveric and clinical randomized studies. Of specific interest to this study is the Transmuscular Quadratus Lumborum(TQL) block, an ultrasound-guided(USG) single-shot nerve block using local anaesthesia, designed to anaesthetize the entire abdominal wall and viscera and the retroperitoneal area. Using ultrasound as visual guidance provides extra safety and insurance of the correct placement of local anaesthetic. The TQL block is described in a recent cadaver study and in several peer review articles. There are two other clinical trials using the TQL-block for percutaneous nefro-lithotripsy and for caesarean section (Eudra-CT 2016-004594-41/2015-004770-16). Both of these trials have ended patient inclusion, and the preliminary data analysis have clearly showed a vast improvement in postoperative pain management and early mobilization with the active TQL blocks - without any adverse events recorded.

The pain from laparoscopic abdominal surgery arises from several locations, both the surgical incisions, the inflation of the entire abdominal wall and parietal peritoneum and traction/stress on the colon.

The innervation of the abdominal wall origins at the ventral rami of the spinal nerves from Th6-L1. The intercostal nerves (VII-XI) and the subcostal nerve all branch out in a lateral and anterior branch. The iliohypogastric and the ilioinguinal nerves innervate the lower part of the abdominal wall. The visceral pain arising from the intraperitoneal organs; i.e. colon, travel via different nerves to join in the thoracic sympathetic trunk before entering the central nervous system. The results from the cadaveric study show a very favourable spread of injectate with the TQL block. Not only does the injected dye in this study spread to colour the ventral rami of the thoracic spinal nerves up to T9 in the thoracic paravertebral space and the iliohypogastric and ilioinguinal nerve; the injectate also spread to colour the thoracic sympathetic trunk. Thus, this seem to indicate that the TQL block can be used to treat not only the pain from the incisions and tears superficially to the colon, but also the pain from the colon itself, and the adjacent intraperitoneal organs and structures, which is affected in patients undergoing laparoscopic hemicolectomy. The cadaveric study has also shown that the lumbar sympathetic trunk and lumbar plexus were not affected by the injected dye. These results seem to imply that there would be minimal or no affection of ambulation or lumbar sympathectomy; i.e. no hypotension or dysfunctional bladder as can often be observed with the epidural technique. Both findings that coincides with the clinical experiences from the investigators pilot studies, and indeed also from the aforementioned clinical trials that have just been finalized.

Cancer progression and the peroperative immunologic stress response:

Studies suggest that events in the perioperative period can induce metastasis formation and tumor growth. Tumor cells are released into the blood stream during surgery and the surgical stress may create a favorable environment for dissemination of tumor cells into distant tissue. This is done by a cascade of pro-cancerous catecholamines, prostaglandins and cytokines combined with an impaired anti-cancerous cell mediated immune response.

Until recently, focus on the anesthetic management of cancer patients has been limited. Relatively small alterations in the perioperative anesthetic management may play a tremendous role in tumor progression. Optimizing anesthesia to reduce the surgical stress response could improve recurrence rates and long-term outcomes for cancer patients by inhibiting perioperative metastasis formation. Regional anesthesia and amide local anesthetics are suspected to calm the immunologic storm of prostaglandins, catecholamines and cytokines when used in the perioperative phase.

Aim: The investigators want to help create an opioid sparing anaesthesia, thus reducing opioid related side effects.

Therefore, the investigators wish to conduct a randomized, controlled and double blind study, comparing the effect of the TQL-block vs. placebo. The aim with this study is to investigate the efficacy of the TQL block vs. placebo in patients undergoing laparoscopic surgery due to colon cancer.

The hypothesis is, that the bilateral TQL block will significantly reduce the opioid consumption during the first 24 postoperative hours and significantly reduce the Numerical Rating Scale (NRS) pain score (0-10) and opioid related side effects.

The investigators will further obtain blood samples in the perioperative period in order to demonstrate effects on the immune system between the two groups. Blood samples and heart rate variability measurement results will be reported in separate peer-review publications.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Scheduled for laparoscopic or robot assisted hemicolectomy or sigmoidectomy due to colon cancer
* Have received thorough information, oral and written, and signed the "Informed Consent" form on participation in the trial
* American Society of Anaesthesiologist physical status classification, class 1-3

Exclusion Criteria:

* Inability to cooperate
* Inability to speak and understand Danish
* Allergy to local anaesthetics or opioids
* Daily intake of opioids (evaluated by the investigators)
* Drug and/or substance abuse
* Local infection at the site of injection or systemic infection
* Difficulty visualisation of muscular and fascial structures in ultrasound visualisation necessary to the block administration
* Pregnant* or breastfeeding
* Daily use of oral or intravenous steroids
* Known immune deficiency (evaluated by the investigators)
* Other simultaneous or previous cancer diagnosis (except non-melanoma skin cancer) within the last five years (within the last five years added 28th nov 2019 after ethics committee approval).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2021-01-03 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | Twenty-four hours postoperative
  Data from PCA pump and patient medical record

SECONDARY OUTCOMES:
Pain during mobilisation | Registered upon arrival at the postanaesthesia care unit (PACU) and again 30 min, 1, 2, 3, 4, 5, 6, 9, 12, 15, 18 and 24 hours postoperative.
  (Numerical rating scale 0-10/10). No pain = 0, worst pain = 10.
Pain at rest | Registered upon arrival at the PACU and again 30 min, 1, 2, 3, 4, 5, 6, 9, 12, 15, 18 and 24 hours postoperative.
  (Numerical rating scale 0-10/10). No pain = 0, worst pain = 10.
An integrated assessment of longitudinally measured pain intensity and opioid consumption | 0-24 hours postoperative
  This assessment is calculated using data from outcome 1 and 2. An individual rank for pain intensity using numerical rating scale (0-10/10), 0-24 hours postoperatively and for total opioid consumption 0-24 hours postoperatively will be combined and compared with a mean rank of all patients (active and placebo). The difference between the individual rank and the mean rank will be expressed as a percentage.
  As described by: Andersen LPK, Gögenur I, Torup H, Rosenberg J, Werner MU. Assessment of Postoperative Analgesic Drug Efficacy: Method of Data Analysis Is Critical. Anesth Analg. 2017 Sep;125(3):1008-13.
Morphine consumption | At 6, 12, 18 postoperative hours.
  Data from PCA pump and patient medical record
Duration of block | Time to first opioid within the first 24 postoperative hours
  How long does the TQL block work
The degree of morphine-related side effects. Nausea or post anaesthesia nausea and vomiting (PONV) registered in the case report form, if any. | 24 hours postoperative
  PONV 0-3; 0=No nausea. 3=Unmanageable nausea
Pain upon ambulation (walking 5 meters with aid) | At 3, 6 and 24 hours postoperative
  Evaluated using Numerical rating scale (0-10/10). No pain = 0, worst pain = 10.
Orthostatic hypotension (yes/no) and orthostatic intolerance i.e. symptoms of orthostatic hypotension without a drop in blood pressure (yes/no). | Before surgery and at 3, 6 and 24 hours postoperative
  Evaluated using standardised test regularly used at the Department of Surgery
Quality of Recovery - 15 questionnaire | Preoperatively and day 1+2 and 10-14 post surgery
  The Quality of Recovery -15 questionnaire results in a score of 0-150. Very poor recovery = 0, excellent recovery = 150. These outcome measures will be correlated with changes in immunologic outcome measures in the perioperative period.
Surgical complications | 30 days post surgery
  Classified using the Clavien-Dindo classification
Time to discharge | 30 days after surgery
  Data from the patient medical record
Heart Rate Variability (HRV) | From block administration and to 24 hours postoperative
  On 24 consecutive patients (3 randomization blocks of 4) data will be obtained on heart rate variability using electrocardiography from block administration and the first 24 hours postoperatively. Minimal changes in HRV characterizes differences in sympathetic stress response between the groups
Whole blood gene expression profiling | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  An evaluation of gene expression fold changes compared to POD 0 using an Affymetrix gene expression array. The investigators will specifically measure relative changes in expression of the GZMB gene, which encodes Granzyme B. Granzyme B is expressed by cytotoxic t-cells and NK-cells. The regularized t-test limma will be used to calculate differences in gene expression between samples taken at different time sets, and the Benjamini Hochberg method using the false discovery rate (FDR) will be used to correct for multiple hypothesis testing.
tumor necrosis factor alpha | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to postoperative day (POD) 0.
interleukin-1b | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to POD 0.
interleukin -2 | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to POD 0.
interleukin-6 | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to POD 0.
interleukin-8 | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to POD 0.
interleukin-10 | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to POD 0.
interleukin-11 | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to POD 0.
interleukin-15 | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to POD 0.
interleukin-17a | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to POD 0.
interleukin-17f | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to POD 0.
interleukin-18 | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to POD 0.
interleukin-22 | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to POD 0.
Granulocyte-macrophage colony-stimulating factor | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of cytokine assays for alterations in inflammation and cancer related immune-function measured by commercial enzyme-linked immunosorbent assays (ELISAs) on a BEP2000 ELISA instrument. Relative changes compared to POD 0.
Hemoglobin | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of standard blood samples that will be obtained and analyzed immediately at each time point. Relative changes compared to POD 0.
Leucocytes including differential count | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of standard blood samples that will be obtained and analyzed immediately at each time point. Relative changes compared to POD 0.
Thrombocytes | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of standard blood samples that will be obtained and analyzed immediately at each time point. Relative changes compared to POD 0.
Alanine aminotransferase (ALAT) | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of standard blood samples that will be obtained and analyzed immediately at each time point. Relative changes compared to POD 0.
Lactate dehydrogenase | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of standard blood samples that will be obtained and analyzed immediately at each time point. Relative changes compared to POD 0.
Bilirubin | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of standard blood samples that will be obtained and analyzed immediately at each time point. Relative changes compared to POD 0.
Prothrombin time (International normalized ratio) | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of standard blood samples that will be obtained and analyzed immediately at each time point. Relative changes compared to POD 0.
Albumin | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of standard blood samples that will be obtained and analyzed immediately at each time point. Relative changes compared to POD 0.
Sodium | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of standard blood samples that will be obtained and analyzed immediately at each time point. Relative changes compared to POD 0.
Potassium | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of standard blood samples that will be obtained and analyzed immediately at each time point. Relative changes compared to POD 0.
C reactive Protein | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of standard blood samples that will be obtained and analyzed immediately at each time point. Relative changes compared to POD 0.
Glucose | Blood samples are taken preoperatively, day 1+2 and 10-14 post surgery
  Part of standard blood samples that will be obtained and analyzed immediately at each time point. Relative changes compared to POD 0.

OTHER OUTCOMES:
Cytokines in LPS stimulated blood | Blood samples are taken preoperatively and day one post surgery
  Difference in cytokine levels (tumor necrosis factor alpha (TNF-a), interleukin-1b (IL-1b), interleukin -2 (IL-2), interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10), interleukin-11 (IL-11), interleukin-15 (IL-15), interleukin-17a (IL-17a), interleukin-17f (IL-17f), interleukin-18 (IL-18), interleukin-22 (IL-22) and GM-CSF, all pg/ml) between postoperative and preoperative whole blood exposed to lipopolysaccharide measured with multiplex assay
Cytokines in CD3+CD28 stimulated blood | Blood samples are taken preoperatively and day one post surgery
  Difference in cytokine levels (tumor necrosis factor alpha (TNF-a), interleukin-1b (IL-1b), interleukin -2 (IL-2), interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10), interleukin-11 (IL-11), interleukin-15 (IL-15), interleukin-17a (IL-17a), interleukin-17f (IL-17f), interleukin-18 (IL-18), interleukin-22 (IL-22) and GM-CSF, all pg/ml)between postoperative and preoperative whole blood exposed to CD3 and CD28 with multiplex assay
Cytokines in Poly I:P stimulated blood | Blood samples are taken preoperatively and day one post surgery
  Difference in cytokine levels (tumor necrosis factor alpha (TNF-a), interleukin-1b (IL-1b), interleukin -2 (IL-2), interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10), interleukin-11 (IL-11), interleukin-15 (IL-15), interleukin-17a (IL-17a), interleukin-17f (IL-17f), interleukin-18 (IL-18), interleukin-22 (IL-22) and GM-CSF, all pg/ml)between postoperative and preoperative whole blood exposed to Polyinosinic:polycytidylic acid with multiplex assay
Cytokines in R848 stimulated blood | Blood samples are taken preoperatively and day one post surgery
  Difference in cytokine levels (tumor necrosis factor alpha (TNF-a), interleukin-1b (IL-1b), interleukin -2 (IL-2), interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10), interleukin-11 (IL-11), interleukin-15 (IL-15), interleukin-17a (IL-17a), interleukin-17f (IL-17f), interleukin-18 (IL-18), interleukin-22 (IL-22) and GM-CSF, all pg/ml)between postoperative and preoperative whole blood exposed to Resiquimod (R848) with multiplex assay

CONTACTS AND LOCATIONS:
Overall Officials: Katrine Tanggaard, MD, Principal Investigator — Department of Anaesthesiology, Zealand University Hospital, Roskilde
Locations (1):
- Zealand University Hospital, Department of Anaesthesiology, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Årsrapporter [Internet]. [cited 2017 Jun 7]. Available from: http://www.dccg.dk/03_Publikation/02_arsraport.html
- [Background] Kehlet H. Postoperative opioid sparing to hasten recovery: what are the issues? Anesthesiology. 2005 Jun;102(6):1083-5. doi: 10.1097/00000542-200506000-00004. No abstract available. PMID 15915017
- [Background] Sondergaard ES, Gogenur I. [Oxidative stress may cause metastatic disease in patients with colorectal cancer]. Ugeskr Laeger. 2015 Apr 27;177(18):857-60. Danish. PMID 26539573
- [Background] Gogenur M, Watt SK, Gogenur I. [Improved immunologic response after laparoscopic versus open colorectal cancer surgery]. Ugeskr Laeger. 2015 Jul 13;177(29):V12140763. Danish. PMID 26239962
- [Background] Sun Y, Li T, Gan TJ. The Effects of Perioperative Regional Anesthesia and Analgesia on Cancer Recurrence and Survival After Oncology Surgery: A Systematic Review and Meta-Analysis. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):589-98. doi: 10.1097/AAP.0000000000000273. PMID 26263074
- [Background] Borglum J, Jensen K, Christensen AF, Hoegberg LC, Johansen SS, Lonnqvist PA, Jansen T. Distribution patterns, dermatomal anesthesia, and ropivacaine serum concentrations after bilateral dual transversus abdominis plane block. Reg Anesth Pain Med. 2012 May-Jun;37(3):294-301. doi: 10.1097/AAP.0b013e31824c20a9. PMID 22476239
- [Background] Borglum J, Maschmann C, Belhage B, Jensen K. Ultrasound-guided bilateral dual transversus abdominis plane block: a new four-point approach. Acta Anaesthesiol Scand. 2011 Jul;55(6):658-63. doi: 10.1111/j.1399-6576.2011.02430.x. Epub 2011 Apr 4. PMID 21463262
- [Background] Jensen K, Baek N, Jensen JT, Brglum J. Bilateral dual transversus abdominis plane block providing surgical anaesthesia for abdominal wall surgery. Anaesthesia. 2013 Jan;68(1):106-8. doi: 10.1111/anae.12103. No abstract available. PMID 23231609
- [Background] Petersen M, Elers J, Borglum J, Belhage B, Mortensen J, Maschmann C. Is pulmonary function affected by bilateral dual transversus abdominis plane block? A randomized, placebo-controlled, double-blind, crossover pilot study in healthy male volunteers. Reg Anesth Pain Med. 2011 Nov-Dec;36(6):568-71. doi: 10.1097/AAP.0b013e3182330b95. PMID 22005660
- [Background] Baerentzen F, Maschmann C, Jensen K, Belhage B, Hensler M, Borglum J. Ultrasound-guided nerve block for inguinal hernia repair: a randomized, controlled, double-blind study. Reg Anesth Pain Med. 2012 Sep-Oct;37(5):502-7. doi: 10.1097/AAP.0b013e31825a3c8a. PMID 22705951
- [Background] Borglum J, Gogenur I, Bendtsen TF. Abdominal wall blocks in adults. Curr Opin Anaesthesiol. 2016 Oct;29(5):638-43. doi: 10.1097/ACO.0000000000000378. PMID 27429253
- [Background] Tanggaard K, Jensen K, Lenz K, Vazin M, Binzer J, Lindberg-Larsen VO, Niegsch M, Bendtsen TF, Jorgensen LN, Borglum J. A randomised controlled trial of bilateral dual transversus abdominis plane blockade for laparoscopic appendicectomy. Anaesthesia. 2015 Dec;70(12):1395-400. doi: 10.1111/anae.13234. Epub 2015 Oct 14. PMID 26464041
- [Background] Børglum J, Moriggl B, Jensen K, Lønnqvist P-A, Christensen AF, Sauter A, et al. Ultrasound-Guided Transmuscular Quadratus Lumborum Blockade. Br J Anaesth [Internet]. 2013 Apr 22 [cited 2017 May 29];111(eLetters Supplement). Available from: https://academic.oup.com/bja/article/doi/10.1093/bja/el_9919/2451466/Ultrasound-Guided-Transmuscular-Quadratus-Lumborum
- [Background] Dam M, Hansen CK, Borglum J, Chan V, Bendtsen TF. A transverse oblique approach to the transmuscular Quadratus Lumborum block. Anaesthesia. 2016 May;71(5):603-4. doi: 10.1111/anae.13453. No abstract available. PMID 27072772
- [Background] Dam M, Moriggl B, Hansen CK, Hoermann R, Bendtsen TF, Borglum J. The Pathway of Injectate Spread With the Transmuscular Quadratus Lumborum Block: A Cadaver Study. Anesth Analg. 2017 Jul;125(1):303-312. doi: 10.1213/ANE.0000000000001922. PMID 28277325
- [Background] Hansen CK, Dam M, Bendtsen TF, Borglum J. Ultrasound-Guided Quadratus Lumborum Blocks: Definition of the Clinical Relevant Endpoint of Injection and the Safest Approach. A A Case Rep. 2016 Jan 15;6(2):39. doi: 10.1213/XAA.0000000000000270. No abstract available. PMID 26771297
- [Background] Mænchen N. Ultrasound-guided Transmuscular Quadratus Lumborum (TQL) Block for Pain Management after Caesarean Section. [cited 2017 May 29]; Available from: https://clinmedjournals.org/articles/ijaa/international-journal-of-anesthetics-and-anesthesiology-ijaa-3-048.php?jid=ijaa
- [Background] Demicheli R, Fornili M, Ambrogi F, Higgins K, Boyd JA, Biganzoli E, Kelsey CR. Recurrence dynamics for non-small-cell lung cancer: effect of surgery on the development of metastases. J Thorac Oncol. 2012 Apr;7(4):723-30. doi: 10.1097/JTO.0b013e31824a9022. PMID 22425921
- [Background] Demicheli R, Biganzoli E, Boracchi P, Greco M, Retsky MW. Recurrence dynamics does not depend on the recurrence site. Breast Cancer Res. 2008;10(5):R83. doi: 10.1186/bcr2152. Epub 2008 Oct 9. PMID 18844974
- [Background] Ciechanowicz SJ, Ma D. Anaesthesia for oncological surgery - can it really influence cancer recurrence? Anaesthesia. 2016 Feb;71(2):127-31. doi: 10.1111/anae.13342. Epub 2015 Dec 16. No abstract available. PMID 26669960
- [Background] Freeman J, Connolly C, Buggy D. Mechanisms of Metastasis of Solid Organ Tumors in the Perioperative Period. Int Anesthesiol Clin. 2016 Fall;54(4):29-47. doi: 10.1097/AIA.0000000000000124. No abstract available. PMID 27648889
- [Background] Horowitz M, Neeman E, Sharon E, Ben-Eliyahu S. Exploiting the critical perioperative period to improve long-term cancer outcomes. Nat Rev Clin Oncol. 2015 Apr;12(4):213-26. doi: 10.1038/nrclinonc.2014.224. Epub 2015 Jan 20. PMID 25601442
- [Background] Yamaguchi K, Takagi Y, Aoki S, Futamura M, Saji S. Significant detection of circulating cancer cells in the blood by reverse transcriptase-polymerase chain reaction during colorectal cancer resection. Ann Surg. 2000 Jul;232(1):58-65. doi: 10.1097/00000658-200007000-00009. PMID 10862196
- [Background] Demicheli R, Retsky MW, Hrushesky WJ, Baum M, Gukas ID. The effects of surgery on tumor growth: a century of investigations. Ann Oncol. 2008 Nov;19(11):1821-8. doi: 10.1093/annonc/mdn386. Epub 2008 Jun 10. PMID 18550576
- [Background] Coffey JC, Wang JH, Smith MJ, Bouchier-Hayes D, Cotter TG, Redmond HP. Excisional surgery for cancer cure: therapy at a cost. Lancet Oncol. 2003 Dec;4(12):760-8. doi: 10.1016/s1470-2045(03)01282-8. PMID 14662433
- [Background] Duff S, Connolly C, Buggy DJ. Adrenergic, Inflammatory, and Immune Function in the Setting of Oncological Surgery: Their Effects on Cancer Progression and the Role of the Anesthetic Technique in their Modulation. Int Anesthesiol Clin. 2016 Fall;54(4):48-57. doi: 10.1097/AIA.0000000000000120. No abstract available. PMID 27648890
- [Background] Bartal I, Melamed R, Greenfeld K, Atzil S, Glasner A, Domankevich V, Naor R, Beilin B, Yardeni IZ, Ben-Eliyahu S. Immune perturbations in patients along the perioperative period: alterations in cell surface markers and leukocyte subtypes before and after surgery. Brain Behav Immun. 2010 Mar;24(3):376-86. doi: 10.1016/j.bbi.2009.02.010. Epub 2009 Feb 28. PMID 19254757
- [Background] Tai LH, de Souza CT, Belanger S, Ly L, Alkayyal AA, Zhang J, Rintoul JL, Ananth AA, Lam T, Breitbach CJ, Falls TJ, Kirn DH, Bell JC, Makrigiannis AP, Auer RA. Preventing postoperative metastatic disease by inhibiting surgery-induced dysfunction in natural killer cells. Cancer Res. 2013 Jan 1;73(1):97-107. doi: 10.1158/0008-5472.CAN-12-1993. Epub 2012 Oct 22. PMID 23090117
- [Background] Zimmitti G, Soliz J, Aloia TA, Gottumukkala V, Cata JP, Tzeng CW, Vauthey JN. Positive Impact of Epidural Analgesia on Oncologic Outcomes in Patients Undergoing Resection of Colorectal Liver Metastases. Ann Surg Oncol. 2016 Mar;23(3):1003-11. doi: 10.1245/s10434-015-4933-1. Epub 2015 Oct 28. PMID 26511261
- [Background] Hiller JG, Hacking MB, Link EK, Wessels KL, Riedel BJ. Perioperative epidural analgesia reduces cancer recurrence after gastro-oesophageal surgery. Acta Anaesthesiol Scand. 2014 Mar;58(3):281-90. doi: 10.1111/aas.12255. Epub 2014 Jan 2. PMID 24383612
- [Background] Gottschalk A, Ford JG, Regelin CC, You J, Mascha EJ, Sessler DI, Durieux ME, Nemergut EC. Association between epidural analgesia and cancer recurrence after colorectal cancer surgery. Anesthesiology. 2010 Jul;113(1):27-34. doi: 10.1097/ALN.0b013e3181de6d0d. PMID 20508494
- [Background] Exadaktylos AK, Buggy DJ, Moriarty DC, Mascha E, Sessler DI. Can anesthetic technique for primary breast cancer surgery affect recurrence or metastasis? Anesthesiology. 2006 Oct;105(4):660-4. doi: 10.1097/00000542-200610000-00008. PMID 17006061
- [Background] Piegeler T, Schlapfer M, Dull RO, Schwartz DE, Borgeat A, Minshall RD, Beck-Schimmer B. Clinically relevant concentrations of lidocaine and ropivacaine inhibit TNFalpha-induced invasion of lung adenocarcinoma cells in vitro by blocking the activation of Akt and focal adhesion kinase. Br J Anaesth. 2015 Nov;115(5):784-91. doi: 10.1093/bja/aev341. PMID 26475807
- [Background] Byrne K, Levins KJ, Buggy DJ. Can anesthetic-analgesic technique during primary cancer surgery affect recurrence or metastasis? Can J Anaesth. 2016 Feb;63(2):184-92. doi: 10.1007/s12630-015-0523-8. PMID 26497721
- [Derived] Balsevicius L, Urbano PCM, Hasselager RP, Mohamud AA, Olausson M, Svraka M, Wahlstrom KL, Oppermann C, Gogenur DS, Holmich ER, Cappelen B, Saekmose SG, Tanggaard K, Litman T, Borglum J, Brix S, Gogenur I. Effect of anterior quadratus lumborum block with ropivacaine on the immune response after laparoscopic surgery in colon cancer: a substudy of a randomized clinical trial. Reg Anesth Pain Med. 2024 Nov 4;49(11):805-814. doi: 10.1136/rapm-2023-104896. PMID 37945063
- [Derived] Tanggaard K, Hasselager RP, Holmich ER, Hansen C, Dam M, Poulsen TD, Baerentzen FO, Eriksen JR, Gogenur I, Borglum J. Anterior quadratus lumborum block does not reduce postoperative opioid consumption following laparoscopic hemicolectomy: a randomized, double-blind, controlled trial in an ERAS setting. Reg Anesth Pain Med. 2023 Jan;48(1):7-13. doi: 10.1136/rapm-2022-103895. Epub 2022 Sep 27. PMID 36167477